CLINICAL TRIAL: NCT04326569
Title: Interest of the Copeptine Dosage in Diagnosis of Post-operative Insipidus Diabetes After Transsphenoidal Pituitary Surgery
Brief Title: Copeptin in the Diagnosis of Post-operative Insipidus Diabetes After Pituitary Surgery
Acronym: Copeptin-surg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA20033
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Pituitary Surgery
Keywords: Pituitary surgery; post-operative insipidus diabetes; copeptin
MeSH Terms: conditions — Diabetes Insipidus | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adults with trans-sphenoidal endoscopic pituitary surgery (Experimental): adult with trans-sphenoidal endoscopic pituitary surgery for tumour of the sellar region
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample to quantify copeptin

SUMMARY:
Endoscopic trans-sphenoidal pituitary endoscopic surgery is one of the main axes of management of tumours of the sellar region.

Central diabetes insipidus is a frequent complication of endoscopic trans-sphenoidal pituitary endoscopic surgery, with a prevalence of up to 30% of cases. It is the consequence of insufficient secretion of the anti-diuretic hormone arginine vasopressin (AVP) by the posterior pituitary (Melmed et al, 2017).

In the absence of specific treatment, diabetes insipidus can lead to severe ionic and osmotic disorders, mainly acute dehydration with the risk of severe consequences particularly neurological.

Monitoring for the appearance of diabetes insipidus is therefore necessary from the immediate post-operative period.

To date, diabetes insipidus is initially suspected before the appearance of major polyuria. Several biological assays (urinary density, natraemia, urinary osmolarity and plasma) can help to confirm the diagnosis, but the sensitivity and specificity of these biomarkers remains quite low for this indication.

The determination of MVA is difficult because this hormone is unstable ex vivo. To date, its use in current practice remains complicated.

MVA and copeptin are derived from the same precursor and are therefore co-secreted by the pituitary gland in equimolar proportions.

Copeptin has a relatively short in vivo half-life of about 25 minutes, as does MVA, but is more stable in vitro when blood has been drawn.

Its use in the early diagnosis of diabetes insipidus after pituitary surgery could therefore be of interest.

DETAILED DESCRIPTION:
Objective is to study the interest of copeptin dosage as an early predictive marker for the diagnosis of post-operatice diabetes insipidus in trans-sphenoidal endoscopic pituitary surgery.

ELIGIBILITY:
inclusion criteria : adult patient patient undergoing pituitary surgery for tumour of the sellar region patient consenting to participate to the study patient enrolled in the national healthcare insurance program

exclusion criteria : Patient with preoperative diabetes insipidus. Patient undergoing pituitary surgery for suspicion of craniopharyngioma Patient undergoing pituitary surgery for pituitary metastases Patient under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Copeptin dosage | Day 1
  Immunoluminometric assay TRACE of the copeptin in pmol/l (Thermofischer)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France